CLINICAL TRIAL: NCT00359567
Title: Comparative Study of Intravenous Single Doses of Palonosetron (PALO) With Granisetron Hydrochloride as a Control in Patients Receiving Highly Emetogenic Chemotherapy
Brief Title: Comparative Study of Palonosetron With Granisetron as a Control in Patients Receiving Highly Emetogenic Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taiho Pharmaceutical Co., Ltd., Taiho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10037030-01
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
Keywords: nausea and vomiting
MeSH Terms: conditions — Vomiting; Nausea | interventions — Palonosetron; Granisetron

ARMS (2):
- 1 (Experimental): palonosetron
  Interventions: Drug: palonosetron
- 2 (Active Comparator): granisetron hydrochloride
  Interventions: Drug: granisetron hydrochloride

INTERVENTIONS:
Drug: palonosetron — intravenous injections of 0.75 mg palonosetron (5 mL) and then granisetron placebo before administration of highly emetogenic chemotherapy, concomitantly administered with corticosteroids.
  Arms: 1
Drug: granisetron hydrochloride — intravenous injections of palonosetron placebo and then 40μg/kg granisetron hydrochloride before administration of highly emetogenic chemotherapy, concomitantly administered with corticosteroids.
  Arms: 2

SUMMARY:
To compare palonosetron with granisetron hydrochloride as a control in the efficacy of intravenous single dose in preventing acute and delayed gastro-intestinal disorders, such as nausea and vomiting induced by highly emetogenic chemotherapy.

DETAILED DESCRIPTION:
This study involves prophylactic single dose of granisetron hydrochloride as a control in the treatment of chemotherapy induced nausea and vomiting (CINV). The primary objective of the study is to verify 0.75 mg palonosetron, concomitantly administered with corticosteroids, is not inferior and superior to granisetron hydrochloride in acute stages 0 - 24 hours and in delayed stages 24 - 120 hours after administration of highly emetogenic chemotherapy, respectively. Corticosteroids are commonly employed in current medical treatments with 5-HT3 receptor antagonists.

This is a multicenter, parallel, group comparative study where subjects are assigned to treatment groups in accordance with a central registration system. After obtaining written informed consent, the patients that satisfy the inclusion criteria without meeting the exclusion criteria are assigned using minimizing procedures to either a single-dose of 0.75 mg palonosetron group or a single-dose of 40 μg/kg granisetron hydrochloride with covariates of chemotherapy regimen, gender and age. A palonosetron group will receive intravenous injections of 0.75 mg palonosetron (5 mL) and then granisetron placebo before administration of highly emetogenic chemotherapy. A granisetron hydrochloride group will be treated with palonosetron placebo and then intravenous 40μg/kg granisetron hydrochloride before administration of highly emetogenic chemotherapy. The onset of nausea and emetic episodes and the time of an antiemetic procedure will be observed for 120 hours after the start of highly emetogenic chemotherapy. The objective is to find the patients' global satisfaction with the antiemetic therapy. Adverse events will also be observed for seven days after the administration of the each drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 or more at the time when they give consent.
* Diagnosed as malignant disease.
* Be naive to chemotherapy or have been treated with single administration of anti-tumor drugs which are classified as low emetogenicity in the first edition of the 2006 NCCN Clinical Practice Guidelines.
* Cisplatin ≥50 mg/m2 Doxorubicin + cyclophosphamide: AC Epirubicin + cyclophosphamide: EC
* WBC ≥ 3000 /mm3 AST < 100 IU/L ALT < 100 IU/L Creatinine clearance ≥ 60 mL/min
* Performance Status : 0 - 2

Exclusion Criteria:

* Severe (requiring hospitalization) and uncontrollable complications.
* Metastases to the brain which are symptomatic.
* Seizure disorder requiring anticonvulsant medication unless clinically stable and free of seizure activity.
* Symptomatic and invasive procedure indicated ascites or pleural effusion.
* Have either gastric outlet stenosis or intestinal obstruction.
* Have ongoing emesis or CTCAE grade 2 or greater nausea.
* QTc > 470 msec in the 12-lead ECG within eight days before registration.
* Known anaphylactic to ingredients of the study drug, namely palonosetron or granisetron hydrochloride injection, or other 5-HT3 receptor antagonists.
* Known anaphylactic to ingredients of dexamethasone.
* Pregnant women, breast-feeding women, or any male or female who are not willing to practice adequate contraception during the study period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1140 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Complete response (CR: no emetic episodes and no rescue medication) rate in acute and delayed nausea and vomiting

SECONDARY OUTCOMES:
Safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Tomohide Tamura, MD, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, 5-1-1 Tsukiji, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Result] Saito M, Aogi K, Sekine I, Yoshizawa H, Yanagita Y, Sakai H, Inoue K, Kitagawa C, Ogura T, Mitsuhashi S. Palonosetron plus dexamethasone versus granisetron plus dexamethasone for prevention of nausea and vomiting during chemotherapy: a double-blind, double-dummy, randomised, comparative phase III trial. Lancet Oncol. 2009 Feb;10(2):115-24. doi: 10.1016/S1470-2045(08)70313-9. Epub 2009 Jan 8. PMID 19135415